CLINICAL TRIAL: NCT01451307
Title: Follow-up Study of Children Aged 2 Years With Gastrointestinal Malformations and Postnatal Surgery
Brief Title: Follow-up of Children With Gastrointestinal Malformations and Postnatal Surgery
Acronym: FraMal
Status: Completed | Type: Observational
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Antje Allendorf-Hofstetter, Principal Investigator, Goethe University
Other Study IDs: 01072011FraMal
Record Dates: First submitted 2011-08-04; First posted 2011-10-13 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Digestive System Abnormalities
Keywords: Congenital abnormalities; Digestive system abnormalities; Neonatal surgery; Neonatal anesthesia; Bayley Scales of Infant Development II
MeSH Terms: conditions — Digestive System Abnormalities; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gastrointestinal malformations: Children who underwent standardized neonatal pediatric surgery due to gastrointestinal malformations
- No gastrointestinal malformations: Control group of healthy children matched concerning gestational age, weight class and gender

SUMMARY:
The aim of this single center study is to measure the impact of standardized neonatal pediatric surgeries due to gastrointestinal malformations on the children's motor and cognitive development and psycho-emotional competence.

To measure the neurodevelopment, the children will be tested with the Bayley Scales of Infant Development II Assessment.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to compare differences in the score of Bayley Scales of Infant Development II Assessment (consisting of cognitive, verbal, nonverbal, motor development levels) between children with gastrointestinal malformations and early postnatal surgery at the age of 2 years and a control group.

The secondary objective is to measure the growth of the patients compared to healthy children in the control group, to capture post-traumatic stress situations in families, and to capture the children's psycho-emotional competence.

Study design:

The study is designed as a cross-sectional single center study. The study patients are children of 2 years of age who underwent neonatal surgery in our clinic since June 2008 due to a gastrointestinal malformation.

The control group consists of matched pairs concerning gestational age, weight and gender.

The study consists of five parts:

* Introductory interview including the medical history
* Bayley Scales of Infant Development II Assessment
* Pediatric examination with anthropometry
* Questionnaire survey of post-traumatic stress situation
* Final conversation with the parents about the results

The neurodevelopmental testing is performed by the child psychologist and the pediatric examination by the pediatrician.

Study population:

The study is purely exploratory and based on the number of patients born in our hospital with the malformations mentioned above (approximately 40).

Each patient is compared against a healthy child of the same gestational age, weight class and gender (control group).

ELIGIBILITY:
Inclusion Criteria:

Patients:

* At follow-up between 18 and 36 months of age
* At birth a gastrointestinal malformation
* Postnatal surgery
* No other serious malformations
* No serious complications of birth (e.g. asphyxia)
* > = 33. week of gestation at birth
* Follow-up appointment when not acutely ill
* Parental Consent

Healthy individuals:

* At follow-up between 18 and 36 months of age
* Uncomplicated postnatal period
* No malformations
* No surgery until follow-up appointment
* > = 33. week of gestation at birth
* Follow-up appointment when not acutely ill
* Parental consent

Exclusion Criteria (both groups):

* Absence of parental consent

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study is purely exploratory and based on the number of patients born in our hospital with the malformations mentioned above (approximately 40).
  Each patient is compared against a healthy child of the same gestational age, weight class and gender (control group).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Score of Bayley Scales of Infant Development II Assessment | 18 Months to 36 Months
  Score consisting of cognitive, verbal, nonverbal and motor development levels

SECONDARY OUTCOMES:
Anthropometric and psychological changes | 18 Months to 36 Months
  * Growth of patients compared to a healthy control group
  * Post-traumatic stress situations in families
  * Psycho-emotional competence of the children

CONTACTS AND LOCATIONS:
Overall Officials: Antje Allendorf-Hofstetter, MD, Principal Investigator — Johann Wolfgang Goethe University Hospital Frankfurt/M, Department of Neonatology
Locations (1):
- Johann Wolfgang Goethe University Hospital, Department of Neonatology, Frankfurt/M, Hesse, Germany

REFERENCES:
- [Background] Walker K, Halliday R, Holland AJ, Karskens C, Badawi N. Early developmental outcome of infants with infantile hypertrophic pyloric stenosis. J Pediatr Surg. 2010 Dec;45(12):2369-72. doi: 10.1016/j.jpedsurg.2010.08.035. PMID 21129547